CLINICAL TRIAL: NCT06393920
Title: PulseSelect PFA Global Registry, a Part of the Medtronic Cardiac Ablation Post-Market Study Platform
Brief Title: PulseSelect™ PFA Global Registry
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PulseSelect™ PFA Registry
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

SUMMARY:
The PulseSelect™ PFA Global Registry is a prospective, global, multi-center, observational post-approval study. Subjects will be treated with the PulseSelect™ PFA System and followed according to SOC.

DETAILED DESCRIPTION:
The PulseSelect™ PFA Global Registry is a prospective, global, multi-center, observational post-market registry. The purpose of this clinical study is to collect clinical performance and safety data in a broad patient population treated with the PulseSelect™ PFA system. The PulseSelect™ PFA System used in the study is market approved. The ablation procedure will be performed according to routine hospital practice. The follow up period is intended to align with standard practice and subjects will be followed for a minimum of 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age or minimum age as required by local regulations.
* Subject has been diagnosed with atrial fibrillation (AF)
* Planned procedure using commercially available PulseSelect™ PFA System.
* Willing to comply with study requirements and give informed consent (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements.

Exclusion Criteria:

* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the global study manager.
* Subject with exclusion criteria required by local law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older with a planned procedure using commercially available PulseSelect™ PFA System
Sampling Method: Non-Probability Sample
Enrollment: 1950 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy-Freedom from Atrial Fibrillation | ≥ 91 days after the index ablation procedure
  Estimate the freedom from AF/AFL/AT recurrence following ablation using the PulseSelect™ PFA system.
Safety- Freedom from Device/Procedure Related Adverse Events | Within 6 months post-ablation
  Estimate serious device and serious procedure-related adverse events for the PulseSelect™ PFA system

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic CAS Chief Medical Officer
Locations (28):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - McGill University Health Centre (MUHC), Montreal, Quebec
- China (5):
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Nanjing Drum Tower Hospital, Nanjing
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Wuhan Asia General Hospital, Wuhan
- France (4):
  - Centre Hospitalier Universitaire de Grenoble - Site Nord, Grenoble
  - Les Hôpitaux de Chartres - Hôpital Louis Pasteur, Le Coudray
  - Hôpital Privé Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Germany (4):
  - Universitäts Klinikum Frankfurt - Goethe-Universität, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Vincenz Krakenhaus Paderborn, Paderborn
  - St. Vincenz-Krankenhaus Paderborn, Paderborn
- Bioclinic Athens, Athens, Greece
- Italy (2):
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Azienda Ospedaliera di Ancona, Ancona
- St Antonius Ziekenhuis, Nieuwegein, Netherlands
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
- Spain (3):
  - Hospital Universitario Reina Sofía, Córdoba
  - H. Univ. Virgen de la Victoria - Malaga, Málaga
  - Complejo Asistencial Universitario de Salamanca, Salamanca
- United Kingdom (2):
  - Basildon and Thurrock University Hospitals, Basildon
  - University Hospitals Coventry & Warwickshire, Coventry